CLINICAL TRIAL: NCT03815617
Title: The Beneficial Effects of a Novel Formulation of Bifidobacterium Longum BB536 and Lactobacillus Rhamnosus HN001 With Vitamin B6 on Gut Microbiota and Intestinal Permeability in IBS Patients.
Brief Title: A Novel Formulation of Bifidobacterium Longum BB536 and Lactobacillus Rhamnosus HN001 With Vitamin B6 on IBS Patients
Acronym: LLB
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, piero portincasa, Principal Investigator, University of Bari
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4651
Record Dates: First submitted 2019-01-22; First posted 2019-01-24 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Intervention Model Description: Patients entered the following program:
  * A run-in period of one month when symptoms, intestinal permeability, intestinal microbiota, and dietary evaluations were performed;
  * Phase 1: randomization to treatment or placebo lasting 30 days;
  * Wash-out period lasting 15 days, at the end of which symptoms were assessed;
  * Phase 2: switch to next treatment in a crossover fashion. Treatment lasted for 30 days and at the end symptoms, intestinal permeability, and intestinal microbiota were evaluated again.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Active Comparator): The study design is a crossover randomized double-blind two-block placebo-controlled single center trial with an allocation ratio of 1:1 conducted between February 2017 and May 2018. Subjects are randomized at baseline visit to receive Block 1 (Zircombi 3 g, containing Bifidobacterium longum BB536 four billion CFU, Lactobacillus rhamnosus HN001 one billion CFU with B6 vitamin 1.4 mg) and Block 2 (placebo: maltodextrins, corn starch, silicon dioxide) depending on the randomization sequence. Subjects received one sachet pack daily containing placebo or probiotic. The active treatment was undistinguishable from placebo by physical and organoleptic characteristics. Participants in the study followed a free diet.
  Interventions: Dietary Supplement: Zircombi
- Placebo (Placebo Comparator): Same appearance of probiotic.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Zircombi — Twenty-five IBS patients (Rome IV criteria) (M:F= 8:17; age 48 yrs ± 11 SD) were enrolled and randomized to treatment or placebo in a a crossover randomized double-blind two-block placebo-controlled trial. Abdominal pain and bloating, intestinal habits, severity of disease, intestinal permeability, and intestinal microbiota were performed at the different time points.
  Arms: Probiotic
Dietary Supplement: Placebo — Given as comparable packets. Same duration.
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) is one of the most frequent functional gastrointestinal disorder with a prevalence ranging from 10 to 15 percent. IBS results from an interaction among several factors, including genetic predisposition, gastrointestinal motility, visceral hypersensitivity, immune activation with minimal inflammation, alterations in intestinal microbiota, increased intestinal permeability, and food sensitivity. Of note, the management of patients with IBS is critical. Since quantitative and qualitative disturbances of intestinal microbiota can occur in IBS, interesting data support the use of probiotics to modulate intestinal microbiota. The present study aimed to investigate the effects of a novel formulation of B. longum BB536 and L. rhamnosus HN001 with vitamin B6 on the gut microbiota and intestinal permeability in IBS subjects.

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) is one of the most frequent functional gastrointestinal disorder with a prevalence ranging from 10 to 15 percent. It is characterized by recurrent chronic abdominal pain or discomfort in the absence of detectable organic causes with two or more of the following conditions: onset associated with a change in frequency of stool, onset associated with a change in form (appearance) of stool, or improvement with defecation.

IBS results from an interaction among several factors, including genetic predisposition, gastrointestinal motility, visceral hypersensitivity, immune activation with minimal inflammation, alterations in intestinal microbiota, increased intestinal permeability, and food sensitivity.

IBS is associated with a high economic burden for the health care costs and work absenteeism.

The disease course is represented by unchanged symptoms in 30 to 50 percent or progression of symptoms in 2 to 18 percent. On the other hand, an improvement in symptoms was recorded in 12 to 38 percent of patients.

Of note, the management of patients with IBS is critical. Several therapeutic options have been proposed looking to the underlying pathophysiological mechanisms (i.e., dietary modification, osmotic laxatives, lubiprostone, guanylate cyclase agonists, 5-hydroxytryptamine (serotonin) 4 receptor agonists, antidiarrheal agents, bile acid sequestrants, 5-hydroxytryptamine (serotonin) 3 receptor antagonists, antispasmodic agents, antidepressants, antibiotics, probiotics, behavior modification, anxiolytics, mast cell stabilizer, and fecal transplantation).

Since quantitative and qualitative disturbances of intestinal microbiota can occur in IBS, interesting data support the use of probiotics to modulate intestinal microbiota. The genus Bifidobacterium is one of the most representative member of the intestinal microbiota with large effects on overall gut physiology. Its metabolic activity results from the degradation of oligo-fructose, production of acetate, and promotion of butyrate production by means of cross-feeding. In particular, B. longum has beneficial effects on the immune system, and can be considered a promising candidate for prevention/treatment of immune-mediated inflammatory diseases.

The combination of specific bacterial strains of Lactobacillus with Bifidobacterium species plays an interesting role in reserving the intestinal dysbiosis. The synergic action results in survival on adverse gastrointestinal conditions, adhesion to intestinal mucosa, immunomodulatory activities, and restoration of gut environment.

The present study aimed to investigate the effects of a novel formulation of B. longum BB536 and L. rhamnosus HN001 with vitamin B6 on the gut microbiota and intestinal permeability in IBS subjects.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IBS according to Rome IV Criteria

Exclusion Criteria:

* Diagnosis of structural abnormality of the GI tract
* Inflammatory bowel disorders
* Biliary duct obstructions
* Gallstones
* Abdominal surgery within the previous six months
* Infective diseases
* Drug or alcohol abuse
* Metabolic disturbances
* Mental illness
* Concomitant immunological, haematological or neoplastic disease
* Severe hepatic insufficiency (i.e., Child-Pugh class C)
* Severe heart failure (NYHA class III-IV)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale, ranging from 0 to 100 | Baseline
  For assessing abdominal pain and bloating
Irritable Bowel Syndrome Symptom Severity Score (IBS-SSS) | Baseline
  Developed by Francis et al. (1997), and categorized as follows: remission (score <75), mild (75-175), moderate (175-300) and severe (>300).
Bristol Stool Form Scale (BSFS) | Baseline
  To assess bowel movements, consisting of a self-report instrument for classifying stool form into seven types ranging from "separate hard lumps like nuts" (type 1) to "watery, no solid pieces" (type 7)
MEDSTYLE questionnaire | Baseline
  A custom-designed questionnaire, tested across different ages, and anthropometric groups in health and disease, to measure anthropometric data, medical history, lifestyle and daily intake of foods. Frequency (day, week or month) and portion sizes (small, medium and large, represented by color pictures) of food consumption were estimated by using 35 food items (156 foods).The adherence to a Mediterranean diet was calculated by analyzing nine food categories with a score ranging from 0 point (lowest adherence) to 18 points (highest adherence).
Intestinal permeability | Baseline
  It was assessed by oral administration of four sugar probes, which selectively characterize the permeability from different tracts of the gastrointestinal system. Sucrose (SO) was used as a marker of gastro-duodenal permeability; lactulose (LA) and mannitol (MA) were used as markers of small intestine permeability also as (LA/MA), and sucralose (SU) as marker of
  8 colonic permeability.
Cultivable intestinal microbiota | Baseline
  It was evaluated by faecal samples (5 g) were mixed with 45 mL sterilized physiological solution and homogenized.
Community level catabolic profiles | Baseline
  Biolog Eco microplates (Biolog, Inc., Hayward, CA, USA) were used to estimate the microbial diversity.
Fecal metabolome | Baseline
  Three grams of fecal sample were placed into 10 mL glass vials and added with 10 μL of 4-methyl- 2-pentanol (final concentration of 33 mg/L) as the internal standard.

CONTACTS AND LOCATIONS:
Overall Officials: Piero Portincasa, Principal Investigator — Professor
Locations (1):
- Clinica Medica "A. Murri", Department of Biomedical Sciences & Human Oncology, University of Bari Medical School, Bari, BA, Italy

REFERENCES:
- [Background] Lovell RM, Ford AC. Global prevalence of and risk factors for irritable bowel syndrome: a meta-analysis. Clin Gastroenterol Hepatol. 2012 Jul;10(7):712-721.e4. doi: 10.1016/j.cgh.2012.02.029. Epub 2012 Mar 15. PMID 22426087
- [Background] Mearin F, Lacy BE, Chang L, Chey WD, Lembo AJ, Simren M, Spiller R. Bowel Disorders. Gastroenterology. 2016 Feb 18:S0016-5085(16)00222-5. doi: 10.1053/j.gastro.2016.02.031. Online ahead of print. PMID 27144627
- [Background] Bonfrate L, Tack J, Grattagliano I, Cuomo R, Portincasa P. Microbiota in health and irritable bowel syndrome: current knowledge, perspectives and therapeutic options. Scand J Gastroenterol. 2013 Sep;48(9):995-1009. doi: 10.3109/00365521.2013.799220. PMID 23964766
- [Background] Camilleri M. Peripheral mechanisms in irritable bowel syndrome. N Engl J Med. 2012 Oct 25;367(17):1626-35. doi: 10.1056/NEJMra1207068. No abstract available. PMID 23094724
- [Background] Sandler RS, Everhart JE, Donowitz M, Adams E, Cronin K, Goodman C, Gemmen E, Shah S, Avdic A, Rubin R. The burden of selected digestive diseases in the United States. Gastroenterology. 2002 May;122(5):1500-11. doi: 10.1053/gast.2002.32978. PMID 11984534
- [Background] El-Serag HB, Pilgrim P, Schoenfeld P. Systemic review: Natural history of irritable bowel syndrome. Aliment Pharmacol Ther. 2004 Apr 15;19(8):861-70. doi: 10.1111/j.1365-2036.2004.01929.x. PMID 15080847
- [Background] Hill C, Guarner F, Reid G, Gibson GR, Merenstein DJ, Pot B, Morelli L, Canani RB, Flint HJ, Salminen S, Calder PC, Sanders ME. Expert consensus document. The International Scientific Association for Probiotics and Prebiotics consensus statement on the scope and appropriate use of the term probiotic. Nat Rev Gastroenterol Hepatol. 2014 Aug;11(8):506-14. doi: 10.1038/nrgastro.2014.66. Epub 2014 Jun 10. PMID 24912386
- [Background] Markowiak P, Slizewska K. Effects of Probiotics, Prebiotics, and Synbiotics on Human Health. Nutrients. 2017 Sep 15;9(9):1021. doi: 10.3390/nu9091021. PMID 28914794
- [Background] Milani C, Lugli GA, Duranti S, Turroni F, Mancabelli L, Ferrario C, Mangifesta M, Hevia A, Viappiani A, Scholz M, Arioli S, Sanchez B, Lane J, Ward DV, Hickey R, Mora D, Segata N, Margolles A, van Sinderen D, Ventura M. Bifidobacteria exhibit social behavior through carbohydrate resource sharing in the gut. Sci Rep. 2015 Oct 28;5:15782. doi: 10.1038/srep15782. PMID 26506949
- [Background] Falony G, Vlachou A, Verbrugghe K, De Vuyst L. Cross-feeding between Bifidobacterium longum BB536 and acetate-converting, butyrate-producing colon bacteria during growth on oligofructose. Appl Environ Microbiol. 2006 Dec;72(12):7835-41. doi: 10.1128/AEM.01296-06. Epub 2006 Oct 20. PMID 17056678
- [Background] Rios-Covian D, Gueimonde M, Duncan SH, Flint HJ, de los Reyes-Gavilan CG. Enhanced butyrate formation by cross-feeding between Faecalibacterium prausnitzii and Bifidobacterium adolescentis. FEMS Microbiol Lett. 2015 Nov;362(21):fnv176. doi: 10.1093/femsle/fnv176. Epub 2015 Sep 28. PMID 26420851
- [Background] Khailova L, Petrie B, Baird CH, Dominguez Rieg JA, Wischmeyer PE. Lactobacillus rhamnosus GG and Bifidobacterium longum attenuate lung injury and inflammatory response in experimental sepsis. PLoS One. 2014 May 15;9(5):e97861. doi: 10.1371/journal.pone.0097861. eCollection 2014. PMID 24830455
- [Background] Toscano M, De Grandi R, Stronati L, De Vecchi E, Drago L. Effect of Lactobacillus rhamnosus HN001 and Bifidobacterium longum BB536 on the healthy gut microbiota composition at phyla and species level: A preliminary study. World J Gastroenterol. 2017 Apr 21;23(15):2696-2704. doi: 10.3748/wjg.v23.i15.2696. PMID 28487606